CLINICAL TRIAL: NCT02754063
Title: Impact of Early Optimization of Brain Oxygenation on Neurological Outcome After Severe Traumatic Brain Injury
Acronym: OXY-TC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 38RC14.039
Record Dates: First submitted 2016-04-15; First posted 2016-04-28 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ICP Management (Active Comparator)
  Interventions: Other: No PbtO2 probes
- PbtO2 + ICP Management (Experimental)
  Interventions: Device: PbtO2 probes

INTERVENTIONS:
Device: PbtO2 probes — PbtO2/ICP/CPP-directed therapy according to international recommendations
  Arms: PbtO2 + ICP Management
Other: No PbtO2 probes — ICP/CPP-directed therapy according to international recommendations
  Arms: ICP Management

SUMMARY:
Post-traumatic brain hypoxia/ischemia develops hours after traumatic brain injury (TBI), and its intensity is directly related to the neurological outcome. The thresholds for irreversible tissue damage following TBI indicate a particular vulnerability of injured brain. Improving brain oxygenation after severe TBI is the focus of modern TBI management in the intensive care unit (ICU).

The calculation of cerebral perfusion pressure (CPP), with CPP = mean arterial pressure (MAP) - intracranial pressure (ICP), has become the most used estimator of cerebral blow flow. To prevent ischemia due to elevated ICP, current international guidelines recommend maintaining CPP at 60-70 mmHg and ICP below 20 mmHg. However, episodes of brain hypoxia/ischemia, as assessed with brain tissue oxygen pressure (PbtO2) measurements, might occur despite optimization of CPP and ICP, and have been independently associated with poorer patient outcome. PbtO2 values lower than 15 mmHg for more than 30 minutes were shown to be an independent predictor of unfavorable outcome and death. The aggressive treatment of low PbtO2 was associated with improved outcome compared to standard ICP/CPP-directed therapy in cohort studies of severely head-injured patients. On the basis of these findings, it is hypothesized that an early optimization of brain oxygenation, together with keeping ICP and CPP within recommended values, could reduce the volume of vulnerable lesions following severe TBI and possibly improve neurological outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75
* Severe non- penetrating TBI (GCS score 3-8) with motor Glasgow score between 1 and 5
* Possible associated extracranial lesions, except tetraplegia
* Initiation of cerebral monitoring within the first 16 hours since primary traumaticinjury
* Indication of ICP monitoring on admission as part of the management
* Indication of continuous sedation/analgesia for more than 48 hours
* Under mechanical ventilation with stable conditions: PaO2//FiO2 over 150 and PaCO2 between 35 and 45 mmHg, mean arterial pressure over 70 mmHg
* Written informed consent from legal surrogate, patient's relative or investigator decision
* Affiliation to the French Social Security or affiliated to a social security system of EU member state, Norway, Lichtenstein, Iceland or Switzerland
* French-speaking or English-speaking patient

Exclusion Criteria:

* Penetrating TBI
* GCS 3 with bilateral fixed dilated pupils
* Decompressive craniectomy and no repositioning of the bone flap after subdural hematoma evacuation surgery prior to enrolment
* Contraindication of ICP and/or PbtO2 monitoring, i.e., hemostasis disorders and brain tissue infection
* Persistent hemodynamic or respiratory instability despite treatments, i.e., mean arterial pressure < 70 mmHg, PaO2/FiO2 <150, PaCO2 <30 mmHg or >45 mmHg or lactate >5 mmol/l if available.
* Hypothermia <34°C at randomization
* Life expectancy < 24 hours
* Cardiac arrest at initial presentation
* Tetraplegia
* Neuropsychiatric co-morbidities that could interfere with 6 and 12-months assessment outcomes.
* Consent refusal
* Pregnancy
* Participation in another therapeutic study with written consent
* Inability to have a 6-months follow-up
* Ischemic stroke after carotid arterial dissection
* Incapacitated patients in accordance with article L 1121-5 to L1121-8 of the public health code.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2021-10-17 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Neurological outcome according to the extended Glasgow Outcome Scale (GOSE) blind assessed | at 6 months post-trauma

SECONDARY OUTCOMES:
Neurological outcome according to the extended Glasgow Outcome Scale (GOSE) and Disability Rating Scale | at 12 months post-trauma (GOSE)
Disability Rating Scale (DRS) | at 6 and 12 months post-trauma
Quality of life assessment: Functional Independence Measure (FIM) and Medical Outcomes Study Short-Form 12 (SF-12) | at 6 and 12 months post-trauma
Mortality rate | at day 28
Therapeutic intensity as reflected by the number of level 2 and level 3 treatments to treat elevated ICP | during the first 5 days of the ICU stay
Incidence of critical events as defined by: ICP >30 mmHg during 30 min at least ICP >40 mmHg during 5 min at least PbtO2 <10 mmHg during 30 min at least (PbtO2 group) | during the first 5 days of the ICU stay

OTHER OUTCOMES:
Ancillary outcome : Volume of cerebral lesions with abnormal MD values, i.e., decreased or increased MD values, using diffusion tensor MR imaging | at day 6-10 following initiation of cerebral monitoring after severe TBI

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François PAYEN, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (26):
- France (26):
  - CHU Angers, Angers
  - General Hospital of Annecy, Annecy
  - University Hospital Besançon, Besançon
  - University Hospital of Bordeaux, Bordeaux
  - CHU CAEN, Caen
  - University Hospital of Clermont-Ferrand, Clermont-Ferrand
  - University Hospital of Dijon, Dijon
  - Grenoble University Hospital, Grenoble
  - University Hospital of Kremlin-Bicetre, Le Kremlin-Bicêtre
  - University Hospital of Lille, Lille
  - University Hospital of Lyon, Lyon
  - University Hospital of Marseille-Nord, Marseille
  - University Hospital of Marseille-Timone, Marseille
  - University Hospital of Montpellier, Montpellier
  - University Hospital of Nancy, Nancy
  - University Hospital of Nice, Nice
  - University Hospital of Nimes, Nîmes
  - University Hospital of Paris-Salpetriere, Paris
  - University Hospital of Poitiers, Poitiers
  - University Hospital of Rennes, Rennes
  - University Hospital of Rouen, Rouen
  - University Hospital of St-Etienne, Saint-Etienne
  - University Hospital Sud Réunion, Saint-Pierre
  - University Hospital of Strasbourg, Strasbourg
  - Hôpital d'Instruction des Armées, Toulon
  - University Hospital of Toulouse, Toulouse

REFERENCES:
- [Background] Cunningham AS, Salvador R, Coles JP, Chatfield DA, Bradley PG, Johnston AJ, Steiner LA, Fryer TD, Aigbirhio FI, Smielewski P, Williams GB, Carpenter TA, Gillard JH, Pickard JD, Menon DK. Physiological thresholds for irreversible tissue damage in contusional regions following traumatic brain injury. Brain. 2005 Aug;128(Pt 8):1931-42. doi: 10.1093/brain/awh536. Epub 2005 May 11. PMID 15888537
- [Background] Brain Trauma Foundation; American Association of Neurological Surgeons; Congress of Neurological Surgeons; Joint Section on Neurotrauma and Critical Care, AANS/CNS; Bratton SL, Chestnut RM, Ghajar J, McConnell Hammond FF, Harris OA, Hartl R, Manley GT, Nemecek A, Newell DW, Rosenthal G, Schouten J, Shutter L, Timmons SD, Ullman JS, Videtta W, Wilberger JE, Wright DW. Guidelines for the management of severe traumatic brain injury. IX. Cerebral perfusion thresholds. J Neurotrauma. 2007;24 Suppl 1:S59-64. doi: 10.1089/neu.2007.9987. No abstract available. PMID 17511547
- [Background] Oddo M, Levine JM, Mackenzie L, Frangos S, Feihl F, Kasner SE, Katsnelson M, Pukenas B, Macmurtrie E, Maloney-Wilensky E, Kofke WA, LeRoux PD. Brain hypoxia is associated with short-term outcome after severe traumatic brain injury independently of intracranial hypertension and low cerebral perfusion pressure. Neurosurgery. 2011 Nov;69(5):1037-45; discussion 1045. doi: 10.1227/NEU.0b013e3182287ca7. PMID 21673608
- [Background] van den Brink WA, van Santbrink H, Steyerberg EW, Avezaat CJ, Suazo JA, Hogesteeger C, Jansen WJ, Kloos LM, Vermeulen J, Maas AI. Brain oxygen tension in severe head injury. Neurosurgery. 2000 Apr;46(4):868-76; discussion 876-8. doi: 10.1097/00006123-200004000-00018. PMID 10764260
- [Background] Stiefel MF, Spiotta A, Gracias VH, Garuffe AM, Guillamondegui O, Maloney-Wilensky E, Bloom S, Grady MS, LeRoux PD. Reduced mortality rate in patients with severe traumatic brain injury treated with brain tissue oxygen monitoring. J Neurosurg. 2005 Nov;103(5):805-11. doi: 10.3171/jns.2005.103.5.0805. PMID 16304983
- [Background] Narotam PK, Morrison JF, Nathoo N. Brain tissue oxygen monitoring in traumatic brain injury and major trauma: outcome analysis of a brain tissue oxygen-directed therapy. J Neurosurg. 2009 Oct;111(4):672-82. doi: 10.3171/2009.4.JNS081150. PMID 19463048
- [Derived] Payen JF, Vilotitch A, Gauss T, Adolle A, Bosson JL, Bouzat P; OXY-TC trial collaborators. Sex Differences in Neurological Outcome at 6 and 12 Months Following Severe Traumatic Brain Injury. An Observational Analysis of the OXY-TC Trial. J Neurotrauma. 2025 Jun;42(11-12):974-984. doi: 10.1089/neu.2024.0390. Epub 2025 Jan 23. PMID 39846855
- [Derived] Payen JF, Launey Y, Chabanne R, Gay S, Francony G, Gergele L, Vega E, Montcriol A, Couret D, Cottenceau V, Pili-Floury S, Gakuba C, Hammad E, Audibert G, Pottecher J, Dahyot-Fizelier C, Abdennour L, Gauss T, Richard M, Vilotitch A, Bosson JL, Bouzat P; OXY-TC trial collaborators. Intracranial pressure monitoring with and without brain tissue oxygen pressure monitoring for severe traumatic brain injury in France (OXY-TC): an open-label, randomised controlled superiority trial. Lancet Neurol. 2023 Nov;22(11):1005-1014. doi: 10.1016/S1474-4422(23)00290-9. PMID 37863590
- [Derived] Mistral T, Roca P, Maggia C, Tucholka A, Forbes F, Doyle S, Krainik A, Galanaud D, Schmitt E, Kremer S, Kastler A, Tropres I, Barbier EL, Payen JF, Dojat M. Automated Quantification of Brain Lesion Volume From Post-trauma MR Diffusion-Weighted Images. Front Neurol. 2022 Feb 23;12:740603. doi: 10.3389/fneur.2021.740603. eCollection 2021. PMID 35281992
- [Derived] Payen JF, Richard M, Francony G, Audibert G, Barbier EL, Bruder N, Dahyot-Fizelier C, Geeraerts T, Gergele L, Puybasset L, Vigue B, Skaare K, Bosson JL, Bouzat P. Comparison of strategies for monitoring and treating patients at the early phase of severe traumatic brain injury: the multicentre randomised controlled OXY-TC trial study protocol. BMJ Open. 2020 Aug 20;10(8):e040550. doi: 10.1136/bmjopen-2020-040550. PMID 32820002